CLINICAL TRIAL: NCT00671346
Title: Combined Analyses and Long-term Follow-up in the Two Norwegian Homocysteine-Lowering B-Vitamin Trials NORVIT and WENBIT
Brief Title: NORVIT and WENBIT - Long-term Follow-up
Acronym: NORVITWENBIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Tromso (Other); Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Ottar Kjell Nygård, MD, PhD, Haukeland University Hospital
Other Study IDs: NSD-17895; REK-267.07 (Other: REK vest); DT-08/00230-2/RVB (Other: Datatilsynet); Hdir-08/623- (Other: Helsedirektoratet)
Record Dates: First submitted 2008-04-29; First posted 2008-05-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Cancer; Myocardial Infarction; Cerebrovascular Stroke
Keywords: Cancer; Coronary artery disease; Myocardial infarction; Cerebrovascular stroke; Homocysteine; Vitamin B Complex; Folic acid; Vitamin B12; Vitamin B6; Pyridoxal phosphate; Osteoporotic fractures; Diabetes
MeSH Terms: conditions — Neoplasms; Myocardial Infarction; Stroke; Coronary Artery Disease; Osteoporotic Fractures; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Participants in NORVIT and WENBIT allocated to daily oral treatment with folic acid 0.8 mg and vitamin B12 0.4 mg
- 2: Participants in NORVIT and WENBIT allocated to daily oral treatment with folic acid 0.8 mg, vitamin B12 0.4 mg and B6 40 mg.
- 3: Participants in NORVIT and WENBIT allocated to daily oral treatment with vitamin B6 40 mg.
- 4: Participants in NORVIT and WENBIT allocated to daily oral treatment with placebo

SUMMARY:
Two large homocysteine-lowering B-vitamin intervention trials have been performed in Norway during the period 1998 to 2005, NORVIT and WENBIT. The main objective in these trials was to study the clinical effects of homocysteine-lowering therapy with folic acid and vitamin B12 in patients with established coronary artery disease. Follow-up was terminated for NORVIT on Marc 31st 2004 and for WENBIT October 5th 2005, and none of the two trials proved any protective effect of the B-vitamin intervention on cardiovascular outcomes.

There is so far no data on possible long-term effects following years of such B-vitamin treatment.

Thus, the main objective of the combinded NORVIT-WENBIT study will will be to evaluate the long-term effect of the B-vitamin intervention on incident life-style diseases including cardiovascular disease, diabetes, osteoporotic fractures and cancer.

A secondary object will be the identification of risk phenotypes or genotypes, and if such risk associations are midified by the B-vitamin intervention

DETAILED DESCRIPTION:
The "homocysteine-hypothesis" of vascular disease has attracted considerable interest, as total plasma homocysteine levels can be easily lowered by folic acid and vitamin B12, raising the prospect that cardiovascular disease could be lowered by such B-vitamin supplementation.

Two large B-vitamin intervention trials have been performed in Norway during the period 1998 to 2005, NORVIT and WENBIT, both registered at ClinicalTrials.gov, identifiers NCT00266487 and NCT00354081, respectively. The main objective in these trials was to study the effects of homocysteine-lowering therapy with folic acid and vitamin B12 to reduce the risk of cardiovascular events in patients with established coronary artery disease. The B-vitamin intervention, which included vitamin B6 in a 2x2 factorial design, was identical in the two trials. Follow-up was terminated for NORVIT on March 31st 2004 and for WENBIT October 5th 2005. Results from the NORVIT trial was published April 2006 {Bonaa, 2006} and preliminary results from the WENBIT trial were presented at the annual congress of the European Society of Cardiology September 4th 2007 {Zegers, 2007}. The WENBIT trial is completed and submitted for publication early in year 2008.

So far, none of the B-vitamin intervention trials have shown any statistically significant favourable effect of homocysteine-lowering therapy with folic acid with or without concomitant vitamin B12 on cardiovascular events {Bazzano, 2006}. In NORVIT there was even a trend towards an increased risk of cardiovascular events (myocardial infarctions) in patients receiving the combination of folic acid, vitamin B12 and vitamin B6. This trend was not observed in WENBIT. However, the treatment with folic acid / B12 was associated With a more rapid progression of angiographic coronary atenoses {Løland, 2010}. Thus, the "homocysteine-hypothesis" of vascular disease has been attenuated through the emergence of these negative trial results, whereas a potential harmful effect of the B-vitamin intervention has been revealed.

There is so far no data on possible long-term effects following years of B-vitamin supplementation. By combining analyses and follow-up in the NORVIT and WENBIT cohorts, we will probably have some more answers both considering possible subgroup and long-term effects of the B-vitamin intervention.

Current data indicate that folate prevents cancer, especially breast and colorectal cancer. However, during the last few years several reports have challenged this assumption. Swedish observational studies found increased risk of colorectal cancer at high blood folate levels {Van Guelpen, 2006} and increased risk of prostate cancer at high levels of folate and vitamin B12 {Hultdin, 2005}. In a randomised trial with folic acid versus placebo to prevent colorectal adenomas, one found increased risk of cancer in the group receiving folic acid, especially of prostate cancer {Cole, 2007}. In a long-term follow-up of women taking high doses of folic acid throughout pregnancy one found a doubled risk of deaths attributable to breast cancer {Charles, 2004}. Recently it has been hypothesized that the implementation of folic acid fortification of foods may have been wholly or partly responsible for the observed increase in colorectal cancer rates in the USA and Canada in the mid to late 1990s {Mason, 2007}. This has led to new hypotheses that folate may prevent carcinogenesis but may enhance the growth of established cancer cells {Ulrich, 2007}. The question of possible adverse effects of folic acid supplementation will be of major importance when public health administrations decide whether to implement or enhance programs folic acid fortification of foods.

The effect of the B-vitamin intervention will also be studied in relation to other life-style diseases like diabetes and osteoprosis.

Additionally, the combined NORVIT-WENBIT cohort will used for observational studies evaluating new risk phenotypes or genotypes and their potential effect modification by the B-vitamin interventions.

ELIGIBILITY:
Inclusion Criteria:

* Randomised in the Norwegian Vitamin Trial (NORVIT) or in the Western Norway B-Vitamin Intervention Trial (WENBIT)

Exclusion Criteria:

* Withdrawn consent to participate in study cohort for post-trial observational follow-up

Ages: 27 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for combined analyses consists of the of 3 749 + 3 090 = 6 839 men and women aged 27 - 86 years when randomised in the NORVIT and WENBIT trials between December 1998 and April 2004. All patients in NORVIT were randomised following an acute myocardial infarction, whereas patients in WENBIT were randomised following coronary angiography, of which 85% had stable angina pectoris, 10% had acute myocardial infarction and 5% had unstable angina pectoris at baseline.
Sampling Method: Probability Sample
Enrollment: 6839 (Estimated)
Dates: Start 1998-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Possible effects of B-vitamin treatment on risk of developing cancer during the trial periods (completed by 2004 and 2005) and during post-trial follow-up. | 1998-2014

SECONDARY OUTCOMES:
The possible effects of B-vitamin treatment on major cardiovascular events, all cause mortality and cause specific death during the trial periods (completed by 2004 and 2005) and during post-trial follow-up. | 1998-2014

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Nygård, MD, PhD, Study Chair — Department of Heart Disease, Haukeland University Hospital
Locations (2):
- Norway (2):
  - Department of Heart Disease, Haukeland University Hospital, Bergen
  - University of Tromsø, Tromsø

REFERENCES:
- [Background] Bonaa KH, Njolstad I, Ueland PM, Schirmer H, Tverdal A, Steigen T, Wang H, Nordrehaug JE, Arnesen E, Rasmussen K; NORVIT Trial Investigators. Homocysteine lowering and cardiovascular events after acute myocardial infarction. N Engl J Med. 2006 Apr 13;354(15):1578-88. doi: 10.1056/NEJMoa055227. Epub 2006 Mar 12. PMID 16531614
- [Background] Bazzano LA, Reynolds K, Holder KN, He J. Effect of folic acid supplementation on risk of cardiovascular diseases: a meta-analysis of randomized controlled trials. JAMA. 2006 Dec 13;296(22):2720-6. doi: 10.1001/jama.296.22.2720. PMID 17164458
- [Background] Clarke R, Armitage J, Lewington S, Collins R; B-Vitamin Treatment Trialists' Collaboration. Homocysteine-lowering trials for prevention of vascular disease: protocol for a collaborative meta-analysis. Clin Chem Lab Med. 2007;45(12):1575-81. doi: 10.1515/CCLM.2007.346. PMID 18265450
- [Background] Van Guelpen B, Hultdin J, Johansson I, Hallmans G, Stenling R, Riboli E, Winkvist A, Palmqvist R. Low folate levels may protect against colorectal cancer. Gut. 2006 Oct;55(10):1461-6. doi: 10.1136/gut.2005.085480. Epub 2006 Apr 25. PMID 16638790
- [Background] Hultdin J, Van Guelpen B, Bergh A, Hallmans G, Stattin P. Plasma folate, vitamin B12, and homocysteine and prostate cancer risk: a prospective study. Int J Cancer. 2005 Feb 20;113(5):819-24. doi: 10.1002/ijc.20646. PMID 15499634
- [Background] Cole BF, Baron JA, Sandler RS, Haile RW, Ahnen DJ, Bresalier RS, McKeown-Eyssen G, Summers RW, Rothstein RI, Burke CA, Snover DC, Church TR, Allen JI, Robertson DJ, Beck GJ, Bond JH, Byers T, Mandel JS, Mott LA, Pearson LH, Barry EL, Rees JR, Marcon N, Saibil F, Ueland PM, Greenberg ER; Polyp Prevention Study Group. Folic acid for the prevention of colorectal adenomas: a randomized clinical trial. JAMA. 2007 Jun 6;297(21):2351-9. doi: 10.1001/jama.297.21.2351. PMID 17551129
- [Background] Charles D, Ness AR, Campbell D, Davey Smith G, Hall MH. Taking folate in pregnancy and risk of maternal breast cancer. BMJ. 2004 Dec 11;329(7479):1375-6. doi: 10.1136/bmj.329.7479.1375. No abstract available. PMID 15591563
- [Background] Mason JB, Dickstein A, Jacques PF, Haggarty P, Selhub J, Dallal G, Rosenberg IH. A temporal association between folic acid fortification and an increase in colorectal cancer rates may be illuminating important biological principles: a hypothesis. Cancer Epidemiol Biomarkers Prev. 2007 Jul;16(7):1325-9. doi: 10.1158/1055-9965.EPI-07-0329. PMID 17626997
- [Background] Ulrich CM, Potter JD. Folate and cancer--timing is everything. JAMA. 2007 Jun 6;297(21):2408-9. doi: 10.1001/jama.297.21.2408. No abstract available. PMID 17551134
- [Background] Ebbing M, Bleie O, Ueland PM, Nordrehaug JE, Nilsen DW, Vollset SE, Refsum H, Pedersen EK, Nygard O. Mortality and cardiovascular events in patients treated with homocysteine-lowering B vitamins after coronary angiography: a randomized controlled trial. JAMA. 2008 Aug 20;300(7):795-804. doi: 10.1001/jama.300.7.795. PMID 18714059
- [Result] Ebbing M, Bonaa KH, Nygard O, Arnesen E, Ueland PM, Nordrehaug JE, Rasmussen K, Njolstad I, Refsum H, Nilsen DW, Tverdal A, Meyer K, Vollset SE. Cancer incidence and mortality after treatment with folic acid and vitamin B12. JAMA. 2009 Nov 18;302(19):2119-26. doi: 10.1001/jama.2009.1622. PMID 19920236
- [Result] Ulvik A, Ebbing M, Hustad S, Midttun O, Nygard O, Vollset SE, Bonaa KH, Nordrehaug JE, Nilsen DW, Schirmer H, Ueland PM. Long- and short-term effects of tobacco smoking on circulating concentrations of B vitamins. Clin Chem. 2010 May;56(5):755-63. doi: 10.1373/clinchem.2009.137513. Epub 2010 Mar 18. PMID 20299681
- [Result] Ebbing M, Bonaa KH, Arnesen E, Ueland PM, Nordrehaug JE, Rasmussen K, Njolstad I, Nilsen DW, Refsum H, Tverdal A, Vollset SE, Schirmer H, Bleie O, Steigen T, Midttun O, Fredriksen A, Pedersen ER, Nygard O. Combined analyses and extended follow-up of two randomized controlled homocysteine-lowering B-vitamin trials. J Intern Med. 2010 Oct;268(4):367-82. doi: 10.1111/j.1365-2796.2010.02259.x. PMID 20698927
- [Derived] Zuo H, Svingen GFT, Tell GS, Ueland PM, Vollset SE, Pedersen ER, Ulvik A, Meyer K, Nordrehaug JE, Nilsen DWT, Bonaa KH, Nygard O. Plasma Concentrations and Dietary Intakes of Choline and Betaine in Association With Atrial Fibrillation Risk: Results From 3 Prospective Cohorts With Different Health Profiles. J Am Heart Assoc. 2018 Apr 12;7(8):e008190. doi: 10.1161/JAHA.117.008190. PMID 29650710
- See also: NORVIT on ClinicalTrials.gov — http://www.clinicaltrials.gov/ct2/results?term=norvit
- See also: WENBIT on ClinicalTrials.gov — http://www.clinicaltrials.gov/ct2/results?term=wenbit